CLINICAL TRIAL: NCT04196660
Title: THE EFFECT OF LABOR DANCE ON THE LABOR PAIN, BIRTH SATISFACTION, NEWBORN APGAR SCORE AND OXYGEN SATURATION LEVEL
Brief Title: THE EFFECT OF LABOR DANCE ON THE LABOR PAIN, BIRTH SATISFACTION AND NEONATAL OUTCOMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Bihter Akın, Asisstant Prof. Dr., Selcuk University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24.03.17/ 17-3/8
Record Dates: First submitted 2019-12-04; First posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Labor Pain; Satisfaction; Infant Conditions
MeSH Terms: conditions — Labor Pain; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: The study sample included 160 pregnant women who had the following characteristics: i) those who were admitted to the Ministry of Health Urla State Hospital for labor ii) those who met the inclusion criteria, and iii) those who had received labor dance training by attending Prenatal Training with their spouses/partners in the prenatal period. The Dance Practitioner Spouse/Partner Group (DPSG) (Experimental) included 40 pregnant women who signed the Informed Consent Form, the Dance Practitioner Midwife Group (DPMG) included 40 pregnant women and midwives who had received labor dance training, and the Control Group included 80 pregnant women who were subjected to routine treatment without dance. The sample size was calculated using a power analysis. The optimum sample size was found to be 160 as Type 1 error α = 0.05 and Type 2 error β = 0.2 (power = 80%).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The Dance Practitioner Spouse/Partner Group (Experimental): The Dance Practitioner Spouse/Partner Group (DPSG)
  Interventions: Behavioral: Labor Dance
- The Dance Practitioner Midwife Group (Experimental): The Dance Practitioner Midwife Group (DPMG) included 40 pregnant women and midwives who had received labor dance training
  Interventions: Behavioral: Labor Dance
- The Control Group (No Intervention): The Control Group included 80 pregnant women who were subjected to routine treatment without dance

INTERVENTIONS:
Behavioral: Labor Dance — The pregnant women and their spouses were trained about the labor dance in the prenatal training without disclosing any information regarding the delivery and labor pain. The pregnant women and their spouses/partners who wanted to perform the practice were asked to inform the researcher when the labor started. The researcher stayed with the pregnant women and their spouses during the practice and labor process. The pregnant women started to dance with their spouses during the active phase of the labor process accompanied by meditation music (on a YouTube channel named Ohgertam Jugrefem) in a dim, silent environment. The spouse or partner massaged the pregnant woman's sacral area while dancing. During the active phase of labor, the pregnant women in the DPMG danced with the midwives who were attendant in the delivery room and who were monitoring the pregnant women's status.
  Arms: The Dance Practitioner Midwife Group; The Dance Practitioner Spouse/Partner Group

SUMMARY:
Objective: This research was conducted to determine the effects of labor dance on perceived birth pain, birth satisfaction, and neonatal outcomes.

Design: This research was an experimental study with three groups. The data were collected during the active phase of labor as three groups; Dance Practitioner Midwife Group (DPMG-40 pregnant), Dancing Practitioner Spouse / Partner Group (DPSG-40 pregnant) and Control Group (CG-80 pregnant).

Setting: This research was conducted at Ministry of Health Izmir Urla State Hospital between April 1, 2017 and October 31, 2017.

Participants: The pregnant women in the DPMG danced with the midwives in charge of the delivery room and following the pregnancy, but those in the DPSG danced with their spouse/partners during the active phase of labor. Labor pains were measured before the labor dance was begun (when the vaginal dilatation was 4 cm) and after the labor dance (when the vaginal dilatation was 9 cm) using a Visual Analogue Scale (VAS). In the postpartum period, the first, fifth, and tenth-minute Apgar scores and oxygen saturation levels of the newborns were measured and recorded. The Mackey Childbirth Satisfaction Rating Scale was applied to evaluate the women's birth satisfaction at the end of the first hour. In the Control Group, only routine practices were implemented in the hospital, and data were collected as indicated in the experimental groups.

DETAILED DESCRIPTION:
During a labor dance, pregnant women's hands were wrapped around the neck of the partner (midwife or spouse), the pregnant woman put her head on her partner's shoulder, and they swung left to right accompanied by calming music. During the labor dance, the partner accompanied the pregnant woman's swinging movements and massaged the pregnant woman's sacral area at the same time. The study showed a positive effect of labor dancing on decreasing birth pain and improving satisfaction and neonatal outcomes whether the dance was performed with the spouse or the midwife during the intrapartum period.

ELIGIBILITY:
Inclusion Criteria:

Those who were admitted to the Ministry of Health Urla State Hospital for labor

* Those whose cervical dilatation between 4 and 8 cm.
* Those who had received labor dance training by attending Prenatal Training with their spouses/partners in perinatal period.
* Those who met the inclusion criteria (Volunteering, term pregnancy (37-41 gestational weeks), single foetus, not having any pregnancy complication (oligohydramniosis and polihydramniosis, placenta previa, pre-eclampsia, premature rupture of membrane, presentation anomalies, intrauterine growth retardation, intrauterine death, macrosomic baby, foetal distress etc.)

Exclusion Criteria:

When delivered by cesarean sectio,

* Labor was inducted
* Narcotic analgesics used

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2017-10-15 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Pregnant women's perceived labor pain | The perceived pain pregnant women in groups were measured and recorded prior to the intervention (when cervical dilatation reached 4-5 cm). This is a 10 cm scale which is labeled "no pain" a
  - A Visual Analogue Scale (VAS) was administered to determine pregnant women's perceived labor pain
pregnant women's satisfaction level | first hour after the delivery
  The Mackey Childbirth Satisfaction Rating Scale was administered in the first hour after
  .the delivery to determine pregnant women's satisfaction level.The Mackey Childbirth. Satisfaction Rating Scale was administered in the first hour after the delivery to determine pregnant women's satisfaction level.Fives likert type consists of 34 items and six sub-dimensions. Bottom dimensions self satisfaction, partner involvement, infant, midwife / nurses, doctors and general satisfaction related questions. The minimum score that can be obtained from the scale is 34 and the highest score is 170.
  The higher the score obtained from the scale, the higher the satisfaction level of women.
Apgar scores | neonatal apgar score was evaluated at the 1st, 5th and 10th minutes after birth. The aim of this study was to evaluate the effects of birth dance on the newborn.
  Newborns' first-minute, fifth-minute, and tenth-minute Apgar scores were evaluated and recorded
oxygen saturation levels | neonatal oxygen saturation level was evaluated at the 1st, 5th and 10th minutes after birth. The aim of this study was to evaluate the effects of birth dance on the newborn.
  Newborns' first-minute, fifth-minute, and tenth-minute oxygen saturation levels were measured on their right hands, and the results were recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) available to other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: December 2019

REFERENCES:
- [Derived] Akin B, Saydam BK. The effect of labor dance on perceived labor pain, birth satisfaction, and neonatal outcomes. Explore (NY). 2020 Sep-Oct;16(5):310-317. doi: 10.1016/j.explore.2020.05.017. Epub 2020 May 30. PMID 32527687